CLINICAL TRIAL: NCT06822296
Title: Effect of Core Stability Training on Segmental Trunk Control and Quality of Life in Children with Spastic Diplegia: a Randomized Controlled Trial
Brief Title: Effect of Core Stability Training on Segmental Trunk Control and Quality of Life in Children with Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Tamer Mohamed El-Saeed, Associate Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004816
Record Dates: First submitted 2024-12-15; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2023-07

CONDITIONS: Spastic Diplegia; Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Core Stability Training (Experimental): receive an experimental intervention in form of functional exercises to improve core
  Interventions: Other: Designed rehabilitation program
- Traditional physical therapy (Active Comparator): Traditional physical therapy used to treat the same condition
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — Exercises to improve function of children with CP
  Arms: Traditional physical therapy
Other: Designed rehabilitation program — Program of exercises to enhance function
  Arms: Core Stability Training

SUMMARY:
Spastic diplegia is a common shape of cerebral palsy that significantly affects trunk control and quality of life in children. Core stability training (CST) has been utilized as a potential intervention to improve the trunk function. This study investigated the effects of CST on segmental trunk control and quality of life in children with spastic diplegia.

Forty children with spastic diplegia (age: 3 - 6 years) were randomly assigned to either a control group (n=20) receiving a selected physical therapy program or an experimental group (n=20) receiving the same program plus a 30-minute CST program three times weekly for 12 weeks. Segmental trunk control was assessed using the Segmental Assessment of Trunk Control (SATCO) scale, and quality of life was measured using the Pediatric Quality of Life Inventory (PedsQL). Both outcome measures were evaluated pre- and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* 3-6 years
* 1 to 1+ spasticity according to modified Ashworth scale
* level II and III according to GMFCs
* able to follow instructions and understand commands

Exclusion Criteria:

* significant visual or auditory problems
* fixed deformities
* Botox injection
* orthopedic surgery

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Segmental Assessment of Trunk Control scale | Baseline and after 12 weeks of training
  Higher scores mean a better outcome. Minimum Score: 0 (No control at any level) Maximum Score: 14 (Full control at all seven levels, each scoring 2)
Quality of Life Inventory Scale | Baseline and after 12 weeks of training
  Higher scores mean a better outcome. Minimum Score: 0 (poorest quality of life) Maximum Score: 100 (best quality of life)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo University, Giza, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Huang C, Chen Y, Chen G, Xie Y, Mo J, Li K, Huang R, Pan G, Cai Y, Zhou L. Efficacy and safety of core stability training on gait of children with cerebral palsy: A protocol for a systematic review and meta-analysis. Medicine (Baltimore). 2020 Jan;99(2):e18609. doi: 10.1097/MD.0000000000018609. PMID 31914039